CLINICAL TRIAL: NCT05092438
Title: An Observational, Retrospective, Clinical Performance Study Testing Residual Specimens of Cerebrospinal Fluid Obtained by Lumbar Puncture From Meningitis/Encephalitis Subjects Using the QIAstat-Dx® Meningitis/Encephalitis Panel
Brief Title: QIAstat-Dx® Meningitis/Encephalitis Panel Performance Evaluation Study 001
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SMF-DHF-18-0489-001
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Meningitis/Encephalitis
MeSH Terms: conditions — Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — frozen residual specimens of CSF obtained by lumbar puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study for performance evaluation of the QIAstat-Dx® Meningitis/Encephalitis Panel in comparison with other chosen comparator methods.

DETAILED DESCRIPTION:
This multicenter study aims to evaluate the performance of QIAstat-Dx Meningitis/Encephalitis (ME) Panel with another validated comparator method.

ELIGIBILITY:
Inclusion Criteria:

* Residual specimens of CSF obtained by lumbar puncture from subjects with signs and symptoms of meningitis and/or encephalitis following completion of routine testing
* Specimen that had not been centrifuged Adequate residual volume (≥400 μl)

Exclusion Criteria:

* Specimens not fitting criteria outlined above
* CSF obtained from an external ventricular drain or shunt source
* Lack of clear subject identification or label on residual banked CSF specimen
* Obvious physical damage of banked residual specimen
* Repeat specimens from the same subject

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects (adults and children) with signs and symptoms of meningitis and/or encephalitis
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
sensitivity | 6 weeks
  positive percentage agreement
specificity | 6 weeks
  negative percentage agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — QIAGEN Gaithersburg, Inc
Locations (1):
- Qiagen, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
all samples are residual and anonymized